CLINICAL TRIAL: NCT02401035
Title: AN OPEN-LABEL, MULTICENTER STUDY TO EVALUATE THE PHARMACOKINETICS OF SINGLE AND MULTIPLE INTRAVENOUS DOSES OF PANTOPRAZOLE IN TWO AGE COHORTS OF HOSPITALIZED PEDIATRIC SUBJECTS 1 TO 16 YEARS OF AGE WHO ARE CANDIDATES FOR ACID SUPPRESSION THERAPY
Brief Title: PREA, PK And Safety PASS Study Of IV Pantoprazole In Pediatric Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated early due to the infeasibility of enrolling the required number of participants per protocol in the 1 <2 years of age cohort.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1791089; 2014-002182-29 (EudraCT Number); B1791089 (Other: Study Number); GERD (Other: Alias Study Number)
Record Dates: First submitted 2014-12-15; First posted 2015-03-27 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: candidate for acid suppression therapy; presumptive diagnosis of GERD; clinical diagnosis of suspected GERD; symptomatic GERD; endoscopically proven GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV pantoprazole (Experimental): Patients will receive 10 mg, 20 mg, or 40 mg IV pantoprazole determined by weight.
  Interventions: Drug: IV pantoprazole

INTERVENTIONS:
Drug: IV pantoprazole — Patients will receive 10 mg, 20 mg, or 40 mg IV pantoprazole determined by weight

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) and safety of intravenous (IV) pantoprazole in patients 1 to 16 years old who are candidates for acid suppression therapy.

DETAILED DESCRIPTION:
In hospitalized pediatric subjects, age 1 to 16 years who in the judgment of the investigator are candidates for acid suppression therapy, the following are the objectives of this trial:

Primary Objectives To characterize the PK of single and multiple IV doses of pantoprazole in pediatric subjects aged 1 to less than 2 years old.

To characterize the PK of single and multiple IV doses of pantoprazole in pediatric subjects aged 2 to 16 years old.

Secondary Objectives To determine the safety, tolerability, and PK of single and multiple IV doses of pantoprazole in each of the independent age cohorts.

To assess the CYP2C19 genotype in pediatric subjects receiving IV pantoprazole, to determine the presence of the gene for the major enzyme responsible for metabolism of pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 1 to 16 years who in the judgment of the investigator are candidates for gastric acid suppression therapy (ie, those with a presumptive diagnosis of GERD, a clinical diagnosis of suspected GERD, symptomatic GERD, or endoscopically proven GERD) and whom the investigator judges would need to receive IV PPI therapy for at least 4 days.
* Body weight > 5th percentile for age.
* Y-site or dedicated IV line for administration of pantoprazole sodium.
* Expected survival for at least 30 days.
* Fertile male and female subjects of childbearing potential at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 28 days after the last dose of assigned treatment. Female subjects of non-childbearing potential must be premenarchal, have undergone hysterectomy with bilateral oophorectomy, have medically confirmed ovarian failure, or achieved post-menopausal status.

Exclusion Criteria:

* Participation in other studies involving investigational drug(s) or treatment with an investigational drug within 30 days or 5 half lives prior to study entry and/or during study participation.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Pregnant females; breastfeeding females; fertile male subjects, and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 28 days after last dose of investigational product.
* Serum CK levels >3x ULN.
* Known history of HIV or clinical manifestations of AIDS.
* Known hypersensitivity to PPIs or to any substituted benzimidazole or to any of the excipients.
* History of treatment with any PPI within 2 days (48 hours) before investigational product dosing on Day 1.
* Use of H2RAs, sucralfate, misoprostol, or prokinetic agents, and bismuth preparations within 1 day (24 hours) before investigational product dosing on Day 1.
* Any disorder requiring chronic (every day) use of warfarin, carbamazepine, or phenytoin, methotrexate, atazanavir or nelfinavir, clopidogrel, and potent inhibitors and inducers of CYP2C19.
* Chronic (daily) use of glucocorticoids. Steroid inhalers and topical steroids may be used.
* Active malignancy of any type, or history of a malignancy (Subject with a history of malignancies that have been surgically removed or eradicated by irradiation or chemotherapy and who have no evidence of recurrence for at least 5 years before Screening are acceptable).
* ALT or BUN >2.0 ULN or estimated creatinine >1.5 X ULN for age or any other laboratory abnormality considered by the Investigator to be clinically significant within 14 days before Screening.
* In the Investigator's opinion, a chronic condition (eg, diabetes, epilepsy), which is either not stable or well controlled and may interfere with the conduct of the study.
* History of sensitivity to heparin or heparin induced thrombocytopenia.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (3):
  - Children's Health Specialty Center Dallas Campus, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital Militar Central "Cirujano Mayor Dr. Cosme Argerich", CABA, Buenos Aires, Argentina
- University clinical center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Georgia (2):
  - JSC Evex Medical Corporation, Tbilisi
  - LTD Imedi Clinic, Tbilisi
- Germany (2):
  - Katholisches Klinikum Bochum, Bochum
  - Zentralapotheke St. Josef-Hospital, Bochum
- Italy (3):
  - Centro Trials - Dipartimento Pediatrico Universitario Ospedaliero Padiglione Salviati, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - IRCCS-Ospedale Pediatrico Bambino Gesù Farmacia Ospedaliera, Roma
- Serbia (2):
  - University Children's Clinic, Belgrade
  - Institute for Child and Youth Health Care of Vojvodina, Novi Sad
- Slovakia (2):
  - Narodny ustav detskych chorob, Bratislava
  - Univerzitna nemocnica Martin, Martin
- Ukraine (3):
  - Komunalne pidpryiemstvo Dnipropetrovskyi spetsializovanyi klinichnyi medychnyi tsentr materi, Dnipro
  - Komunalne nekomertsiine pidpryiemstvo Ivano-Frankivska oblasna dytiacha klinichna likarnia, Ivano-Frankivsk
  - Komunalne nekomertsiine pidpryiemstvo "Khersonska dytiacha oblasna klinichna likarnia", M. Kherson

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1791089

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 19 participants were enrolled. Nineteen participants were randomized and assigned to a study treatment out of which, 1 participant was not randomized to any study treatment.
Groups:
- Cohort 1 (>=1 to < 2 Years): Participants aged greater than or equal to (>=) 1 year to less than (<) 2 years received intravenous pantoprazole sodium as per body weight with maximum dose not exceeded 40 milligrams (mg), once daily for 4 to 7 days, approximately every 24-hours, preferred in the morning.
- Cohort 2 (>=2 to <16 Years): Participants aged >= 2 to < 16 years received intravenous pantoprazole sodium as per body weight with maximum dose not exceeded 40 mg, once daily for 4 to 7 days, approximately every 24-hours, preferred in the morning.
Period: Overall Study
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Started | 3 | 16
Treated | 2 | 16
Completed | 2 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in analysis.
Groups:
- Cohort 1 (>=1 to < 2 Years): Participants aged >= 1 year to < 2 years received intravenous pantoprazole sodium as per body weight with maximum dose not exceeded 40 mg, once daily for 4 to 7 days, approximately every 24-hours, preferred in the morning.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years) | Total
Number analyzed (Participants) | 3 | 16 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.00 (0.000) | 9.31 (4.729) | 8.00 (5.323)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 3 | 9 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 16 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 16 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clearance (CL) of Pantoprazole
Description: Data reported below is combined for Days 1, 2 and 7.
Time Frame: 0.25, 1 to 2, 3 to 4, and 5 to 6 hours post-dose on Day 1; 0.25, 0.5, 1 to 2, 3 to 4, and 5 to 6, 8, and 12 hours post-dose on Day 2; 0.25, 0.5, 1, 2, 4, 8, and 12 hours post-dose on Day 7
Population: The pharmacokinetic (PK) parameter analysis population included all participants treated with pantoprazole who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Liter per hour | 1.930 (82) | 4.739 (71)

2. Primary Outcome: Volume of Distribution (Vd) of Pantoprazole
Description: Data reported below is combined for Days 1, 2 and 7.
Time Frame: as for outcome 1
Population: The PK parameter analysis population included all participants treated with pantoprazole who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Liter | 1.622 (58) | 5.584 (74)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Pantoprazole: Single Dose
Description: The results for Cmax were presented separately for single dose and multiple doses.
Time Frame: 0.25, 1, 2, 3 to 4, and 5 to 6 hours post-dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Nanogram per milliliter (ng/mL) | 5259 (60) | 4280 (48)

4. Secondary Outcome: Cmax of Pantoprazole: Multiple Dose
Description: Data reported below is combined for Days 2 and 7.
Time Frame: 0.25, 0.5, 1 to 2, 3 to 4, and 5 to 6, 8, and 12 hours post-dose on Day 2; 0.25, 0.5, 1, 2, 4, 8, and 12 hours post dose on Day 7
Population: The PK parameter analysis population included all participants treated with pantoprazole who had at least 1 of the PK parameters of primary interest. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 15
ng/mL | 5259 (60) | 4423 (47)

5. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to 24 Hour (AUC24) of Pantoprazole: Single Dose
Description: The results for AUC24 were presented separately for single dose and multiple doses.
Time Frame: 0.25, 1, 2, 3 to 4, and 5 to 6 hours post-dose on Day 1; 24 hours post dose on Day 1 (pre dose on Day 2)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram* hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Nanogram* hour per milliliter (ng*hr/mL) | 6022 (84) | 6533 (62)

6. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to 24 Hour (AUC24) of Pantoprazole: Multiple Dose
Description: Data reported below is combined for Days 2 and 7.
Time Frame: as for outcome 4
Population: The PK parameter analysis population included all participants treated with pantoprazole who had at least 1 of the PK parameters of primary interest. Since dosing interval between 2 doses are 24 hours, individual post-hoc estimated AUC from population PK analysis is AUC24. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 15
ng*hr/mL | 5705 (82) | 6690 (60)

7. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Pantoprazole: Single Dose
Description: The results for AUCinf were presented separately for single dose and multiple doses.
Time Frame: 0.25, 1, 2, 3 to 4, and 5 to 6 hours post-dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
ng*hr/mL | 6022 (84) | 6542 (62)

8. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Pantoprazole: Multiple Dose
Description: Data reported below is combined for Days 2 and 7.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 15
ng*hr/mL | 5708 (82) | 6707 (61)

9. Secondary Outcome: Terminal Half-Life (t1/2) of Pantoprazole
Description: Data reported below is combined for Days 1, 2 and 7.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Hours | 2.805 (0.1909) | 3.767 (0.6802)

10. Secondary Outcome: Number of Participants According to CYP2C19 Genotyping
Description: CYP2C19 genotype was assessed in pediatric participants who received intravenous pantoprazole sodium and determined the presence of the gene for the major enzyme responsible for metabolism of pantoprazole.
Time Frame: Day 1
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant who was administered a product; the event need not necessarily had a causal relationship with the treatment or usage.
Time Frame: From Day 1 up to 34 days after the last dose (maximum up to 41 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 8

12. Secondary Outcome: Number of Participants With Laboratory Abnormalities of Potential Clinical Concern
Description: Number of participants with abnormalities in laboratory parameters of potential clinical concern were reported in this outcome measure. The criteria to determine the abnormalities was determined by the investigator.
Time Frame: Up to Day 9
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Physical Examination Abnormalities of Potential Clinical Concern
Description: Number of participants with abnormalities in physical examination of potential concern were reported in this outcome measure. The criteria to determine the abnormalities was determined by the investigator.
Time Frame: At screening (Day 0)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Blood Pressure Abnormalities of Potential Clinical Concern
Description: Number of participants with abnormalities in blood pressure of potential clinical concern were reported in this outcome measure. The criteria to determine the abnormalities was determined by the investigator.
Time Frame: Up to Day 9
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Pulse Rate Abnormalities of Potential Clinical Concern
Description: Number of participants with abnormalities in pulse rate of potential clinical concern were reported in this outcome measure. The criteria to determine the abnormalities was determined by the investigator.
Time Frame: Up to Day 9
Population: Safety analysis set included all the participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
Number analyzed (Participants) | 2 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to 34 days after the last dose (maximum up to 41 days)
Description: Same event may appear as both serious adverse event (SAE) and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants who received at least 1 dose of study medication.
Arm/Group | Cohort 1 (>=1 to < 2 Years) | Cohort 2 (>=2 to <16 Years)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/16
Other Adverse Events (participants affected / at risk) | 0/2 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (>=1 to < 2 Years) (N=2) | Cohort 2 (>=2 to <16 Years) (N=16)
Rotavirus infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (>=1 to < 2 Years) (N=2) | Cohort 2 (>=2 to <16 Years) (N=16)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Catheter site erythema (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Catheter site pruritus (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Vessel puncture site erythema (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT02401035/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT02401035/SAP_001.pdf